CLINICAL TRIAL: NCT05840263
Title: Developing a Couple-Based Mindfulness Intervention for Metastatic Colorectal Cancer: Qualitative Phase
Brief Title: Couple-Based Mindfulness Intervention for Metastatic Colorectal Cancer
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 22-2246.cc; K08CA267313 (NIH)
Record Dates: First submitted 2023-04-21; First posted 2023-05-03 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Metastatic Colorectal Cancer Patients: We anticipate enrolling up to a total of 18 patients who have been diagnosed with metastatic colorectal cancer; 12 patients will participate in the qualitative interview, and 6 patients will participate in the cognitive interview.
  Interventions: Behavioral: Qualitative interview; Behavioral: Cognitive Interviews
- Metastatic Colorectal Cancer Patients Partners: We anticipate enrolling up to a total of 18 partners of patients who have been diagnosed with metastatic colorectal cancer; 12 partners will participate in the qualitative interview, and 6 paartners will participate in the cognitive interview.
  Interventions: Behavioral: Qualitative interview; Behavioral: Cognitive Interviews
- Clinicians: We anticipate enrolling 12 clinicians (including physicians, nurse practitioners, physician assistants, mental health providers, other advanced practice clinicians) who treat patients with colorectal cancer at the University of Colorado to participate in qualitative interviews. We seek to enroll a variety of clinicians from advanced practiced clinical roles (physicians, nurse practitioners, and mental health providers) to capture diverse perspectives.
  Interventions: Behavioral: Qualitative interview

INTERVENTIONS:
Behavioral: Qualitative interview — Qualitative interviews will cover four main goals including: (1) key sources of distress in mCRC patients and partners; (2) perceptions of mindfulness, including benefits, definitions, and applications; (3) barriers and facilitators of participation (e.g. home-based and couple-based skills practice, enrollment); and (4) session format preferences, such as session length and frequency.
Behavioral: Cognitive Interviews — The objective of the cognitive interviews (60 minutes, led by the PI) is to ensure the comprehensibility and appropriateness of the drafted participant materials. Published guidelines note a sample size of 12 participants (6 mCRC couples) should be sufficient. Participants will be asked to read, review, and mark up the participant materials in order to identify sections that were difficult to understand. They will also be asked to test playing segments of the audio/video recordings to ensure ease of use. A semi-structured interview format will be used to elicit feedback, including a standard verbal survey assessing ease of reading the material, any difficulties experienced, and suggestions they have for improving the ease of material use. Information generated will be used to update materials as necessary.
  Groups: Metastatic Colorectal Cancer Patients; Metastatic Colorectal Cancer Patients Partners

SUMMARY:
The overall objective of this study is to develop a novel couple-based mindfulness intervention aimed at reducing distress in patients with metastatic colorectal cancer (mCRC) and their partners.

DETAILED DESCRIPTION:
The overall objective of this study is to develop a novel couple-based mindfulness intervention aimed at reducing distress in patients with metastatic colorectal cancer (mCRC) and their partners. The intervention is named "MIND-Together" (Mindfully Navigating Distress Together). MIND-Together will be the first mindfulness-based intervention designed to reduce mCRC couples' distress by targeting their unique psychosocial needs. The intervention is projected to be a 4-session intervention delivered by a trained therapist to individual couples facing mCRC (i.e., a patient and his/her intimate partner) via video-conference (e.g., Zoom).

ELIGIBILITY:
Patient Inclusion Criteria:

* Provision to sign and date the consent form.
* Stated willingness to comply with all study procedures and be available for the duration of the study.
* Be aged > 18 years.
* Fluent in English language
* Be a person (i.e., patient) diagnosed with metastatic colorectal cancer (mCRC), a partner (e.g., spouse) of someone diagnosed with mCRC, or a clinician who treats patients diagnosed with mCRC.

Additional patient participant inclusion criteria:

* Has a current diagnosis of metastatic (Stage IV, recurrent) colorectal cancer
* Has an ECOG status <2 or otherwise deemed appropriate for study participation by a clinician
* Is in a committed relationship with a romantic partner for >6 months
* Has access to computer/internet through with video-conferencing (phone, laptop, tablet, desktop computer)
* Indicates a score >0 on the Distress Thermometer

Additional partner participant inclusion criteria:

* Has been in a committed relationship >6 months with a patient who meets the above eligibility criteria
* Has access to computer/internet through with video-conferencing (phone, laptop, tablet, desktop computer)
* Indicates a score >0 on the Distress Thermometer

Additional clinician participant inclusion criteria:

∙Is a physician or advanced practice clinician (e.g., oncologist, nurse practitioner, physician assistant, psychologist, mental health provider, etc.)

Exclusion Criteria:

∙Has a serious mental illness (e.g., psychotic disorder), cognitive impairment (e.g., dementia), or medical condition (e.g., significant impaired sight/hearing) that would compromise participation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Metastatic Colorectal Cancer Patients
  Metastatic Colorectal Cancer Patients' Partners
  Clinicians (including physicians, nurse practitioners, physician assistants, mental health providers, other advanced practice clinicians) who treat patients with colorectal cancer at the University of Colorado to participate in qualitative interviews.
Sampling Method: Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Identify the needs of mCRC patients for intervention content | During the one-time qualitative interview
  Completed through semi-structured qualitative interviews
Identify the preferences of mCRC patients for intervention content | During the one-time qualitative interview
  Completed through semi-structured qualitative interviews
Identify the needs of mCRC patients' partners for intervention content | During the one-time qualitative interview
  Completed through semi-structured qualitative interviews
Identify the preferences of mCRC patients' partners for intervention content | During the one-time qualitative interview
  Completed through semi-structured qualitative interviews
Identify the preferences of mCRC patients for intervention format (eg, session length) | During the one-time qualitative interview
  Completed through semi-structured qualitative interviews
Identify the preferences of mCRC patients' partners for intervention format (eg, session length) | During the one-time qualitative interview
  Completed through semi-structured qualitative interviews
Identify the preferences of mCRC patients partners for intervention format | During the one-time qualitative interview
  Completed through semi-structured qualitative interviews
Extract key themes to integrate into preliminary drafts | During the one-time qualitative interview
  analyze these qualitative data to extract key themes and will integrate the findings with preliminary drafts of the MIND-Together protocol (e.g., participant handouts, therapist manual).

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Zimmaro, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Cancer Center, Aurora, Colorado, United States